CLINICAL TRIAL: NCT06269055
Title: Long-term Result of DTPA Chelation for Gadolinium Deposition Disease
Brief Title: Long-term Result of DTPA (Diethylenetriamine Pentaacetate) Chelation for Gadolinium Deposition Disease
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Lorrin M Koran, MD, Professor of Psychiatry and Behavioral Sciences, Stanford University
Other Study IDs: 73151
Record Dates: First submitted 2024-02-12; First posted 2024-02-21 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-05

CONDITIONS: Gadolinium Deposition Disease; Ca-DTPA
Keywords: DTPA, chelation
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Interview — Telephone interview and questionnaires about the results and side effects experienced
  Other Names: Telephone interview and written questionnaire completion

SUMMARY:
This study is aimed at describing the degree of benefit, if any, and the adverse effects, if any, from receiving 5 or more treatment sessions of Gadolinium Deposition Disease using two-day chelation treatment with the chelating agents Calcium Diethylenetriamine pentaacetate (Ca-DTPA) and Zinc Diethylenetriamine pentaacetate (Zn-DTPA).

DETAILED DESCRIPTION:
Potential participants will be invited to contact Dr. Koran by email to receive a telephone screening Informed Consent. Those who provide informed consent will have their questions about the study answered and their interest and eligibility assessed via telephone interview. Those who wish to participate will be sent an Informed Consent for study participation. Those who return the consent will be sent four study questionnaires for completion and return. The returned forms will be reviewed by Dr. Koran or his co-investigator, and a follow-up phone call will be offered via Secure Stanford email. The phone call will involve answering any new questions the participant has, and clarifying the participant's responses to the data collection forms if clarification is needed. Participants who wish to receive a summary of the study's results once it is completed and accepted for publication, will be emailed a summary via Secure Stanford email.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older,
2. Diagnosis of Gadolinium Deposition Disease (GDD) established by treating MD according to current criteria and confirmed by investigator review of screening questionnaire (dx criteria: presence of at least 3 of 8 symptoms-cognitive disturbance, extremity pain, arthralgia, chest wall pain, skin pain, headache, skin induration, and skin hyperpigmentation; and, had an unprovoked 24-hour Gd urine excretion level exceeding the laboratory norm at least 28 days after the symptom-inducing MRI;
3. has had five or more 2-day chelation treatments with Ca-DTPA/Zn-DTPA;
4. will be at least 2 weeks post the last chelation treatment at the time of completing the patient data-gathering questionnaires.
5. no more than 2 years have elapsed since the last DTPA chelation.

Exclusion Criteria:

1. Not fluent in written and spoken English; 2. having impaired hearing that significantly decreases the person's ability to communicate via telephone; 3. Prisoners; 4. Unable to provide informed consent; 5. Participating or having participated in protocols involving a pharmacological treatment of GDD other than DTPA chelation. Note: brief pre- or post-DTPA chelation to prevent GDD symptom flare is not an exclusion criterion.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in the U.S. who developed Gadolinium Deposition Disease (GDD) within 28 days of undergoing a contrast-assisted MRI, in which the contrast agent contained the metal gadolinium, and who retained enough gadolinium to have abnormally high 24-hour urine levels 28 or more days post MRI. Participants must satisfy the Inclusion/Exclusion criteria noted above.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rating of Gadolinium Deposition Disease Symptoms at start of GDD and currently | Two or more weeks after the last of 5 of more DTPA chelation treatments
  Patient-completed data regarding symptoms experienced and their intensity when they began and currently, rated from 0 (none) to 5 (very severe). Outcome measure will be change in each symptom's intensity.

SECONDARY OUTCOMES:
PROMIS Item Bank v2.0 - Cognitive Function- Short Form 8a | Past 7 days
  An 8-item patient rated questionnaire with ratings of cognitive symptoms from Very Often to Never for each item, rated 5 (Never) to 1 (Very often). Higher scores indicate better cognitive function.
Sheehan Disability Scale | Past week
  A brief, patient-rated measure of disability and impairment in Work/School, Social Life, and Family Life/Home Responsibilities. Each area is rated from 0 (no disability) to 10 (extreme disability). Higher scores indicate greater disability in the life area rated.

OTHER OUTCOMES:
DTPA-chelation side effects form | Onset on the day of or within one day of DTPA chelation
  Checklist form regarding possible side effects of DTPA chelation

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Semelka RC, Ramalho M. Gadolinium Deposition Disease: Current State of Knowledge and Expert Opinion. Invest Radiol. 2023 Aug 1;58(8):523-529. doi: 10.1097/RLI.0000000000000977. Epub 2023 Apr 11. PMID 37058336